CLINICAL TRIAL: NCT03673514
Title: Direct Anterior Versus Posterior Approach for Total Hip Arthroplasty: a Multicentric Prospective Randomized Clinical Study
Brief Title: Anterior vs Posterior Approach in THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Kevin Moerenhout, Orthopedic Surgeon, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CÉR : 2009-09-67;2010-415
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Total Hip Arthroplasty
Keywords: Direct anterior approach; posterior approach
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: However, the decision to discharge subjects was made by physiotherapists blinded to treatment and based on objective criteria. These criteria were: 1) being autonomous for transfer from bed/chair to upright position 2) being able to walk with walking aid 3) climbing stairs in a safe way 4) having a pain level contained by painkillers. No restrictions were recommended for either group. The same rehabilitation and pain protocols were used for both approaches. In addition, statistical analyses were performed by an independent consultant who remained blinded to treatment group assignment.
Oversight: FDA-regulated Drug: No

ARMS (2):
- THA Posterior Approach (Active Comparator): The posterior approach to the hip has been described by many authors and yields good results. Implants used were Quadra®-H stem and Versacup® hip system, Medacta, Switzerland, with metal on polyethylene bearing. All implants were non-cemented.
  Interventions: Procedure: Total hip arthroplasty
- THA Direct anterior approach (Active Comparator): The modified Hueter approach, based on the Smith-Peterson approach, was performed for the direct anterior minimally invasive surgery. This approach could have some advantages as it is a muscle sparing approach, hence yielding a faster recovery. A traction table was used for DAA as surgeons were trained to use this method. No intra-operative fluoroscopy was used for implant confirmation.Implants used were Quadra®-H stem and Versacup® hip system, Medacta, Switzerland, with metal on polyethylene bearing. All implants were non-cemented.
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — Two fellowship-trained surgeons in two separate hospitals performed all procedures. Both surgeons had previously performed over 100 cases with each approach, before initiating this study

SUMMARY:
Determining the best approach for a total hip arthroplasty (THA) implies that the procedure is kind on soft tissues, with the lowest complication rates, and easily reproducible. Although there have been several attempts to resolve this issue in the last decade, a definitive answer has not been found. Therefore, the investigators performed a prospective study to compare direct anterior versus posterior approach based on (1) hospital stay, (2) functional outcome, (3) pain, (4) implant position (5) complications and (6) surgical time.

DETAILED DESCRIPTION:
In this multicentric, prospective, randomized clinical trial, 55 total hip arthroplasties were performed on 50 patients between February 2011 and July 2013. Patients meeting the inclusion criteria underwent surgical treatment using the DAA or PA, according to a randomization process. Radiological analysis assessed implant position, limb lengthening, and potential implant related complications. X-rays were performed at subsequent follow-up visits and consisted of an antero-posterior (AP) pelvic X-ray and a lateral projection of the hip. Two independent observers, not involved with patients or surgeries, reviewed all postoperative radiographs independently.Two fellowship-trained surgeons in two separate hospitals performed all procedures. Both surgeons had previously performed over 100 cases with each approach, before initiating this study.

Patients underwent either the posterior or direct anterior approach.

ELIGIBILITY:
Inclusion Criteria:

* primary total hip replacement due to osteoarthrosis or osteonecrosis
* patients older than 50 years.

Exclusion Criteria:

* inflammatory arthritis,
* any previous ipsilateral hip surgery
* suffering from proximal femoral deformity
* BMI over 40
* active infection
* severe contralateral hip disease, muscle contractures or neuromuscular pathology
* requiring structural bone grafts.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Hospital stay | Between 0 days and 1 month, average of 4 days
  Length in days of hospital stay

SECONDARY OUTCOMES:
functional recovery | 2 weeks, 4 weeks, 3 months, 6 months, 1 year, 2 years and 5 years postoperatively
  The Harris Hip Score (HHS) was used to measure pain and function.Grading for the Harris Hip Score is interpreted on a scale of 0 to 100 as follows: results <70 are Poor; 70 - 79 are Fair; 80-89 are Good; 90 -100 are Excellent
pain assessment: VAS | 2 weeks, 4 weeks, 3 months, 6 months, 1 year, 2 years and 5 years postoperatively
  Visual Analog Scale (VAS) was used. The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases. The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The pain VAS is a single-item scale, anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) . It is one total score, without subscale. As the lowest score of zero means no pain, it is the best possible outcome. As the highest score of 100 means the worst imaginable pain, it is the worst possible outcome.
implant position | 2 weeks, 4 weeks, 3 months, 6 months, 1 year, 2 years and 5 years postoperatively
  Radiological assessment
number of patients with per/post surgical complications. | 2 weeks, 4 weeks, 3 months, 6 months, 1 year, 2 years and 5 years postoperatively
  Possible complications are: peroperative fracture, hip dislocation, infection, neurologic complication, vascular complication or hematoma.
surgical time | Up to 240 minutes
  Surgical time in minutes

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Derived] Moerenhout K, Derome P, Laflamme GY, Leduc S, Gaspard HS, Benoit B. Direct anterior versus posterior approach for total hip arthroplasty: a multicentre, prospective, randomized clinical trial. Can J Surg. 2020 Sep-Oct;63(5):E412-E417. doi: 10.1503/cjs.012019. PMID 33009898